CLINICAL TRIAL: NCT06547242
Title: Bioequivalence Trial of BC-T4CYS 150 µg Tablets Versus Letrox® 150 µg in Healthy Subjects
Brief Title: Levothyroxine-sodium Bioequivalence Trial With Oral Single Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Berlin-Chemie AG Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BCBE/21/BTX-BE/001; 2021-001454-62 (EudraCT Number)
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2022-01

CONDITIONS: Healthy
MeSH Terms: interventions — Thyroxine; Tablets

STUDY DESIGN:
Intervention Model Description: Single centre, open-label, randomised (order of treatments), balanced, 2-period, 2-sequence, single dose cross-over trial with administrations under fasting conditions separated by a washout period of at least 45 treatment-free days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BC-T4CYS 150 µg tablet (Berlin-Chemie AG) (Experimental): BC-T4CYS 150 µg tablet (Berlin-Chemie AG), oral single dose administration of 4 tablets (600 µg levothyroxine-sodium)
  Interventions: Drug: Levothyroxin
- Letrox® 150 µg tablet (Berlin-Chemie AG), (Active Comparator): Letrox® 150 µg tablet (Berlin-Chemie AG), oral single dose administration of 4 tablets (600 µg levothyroxine-sodium)
  Interventions: Drug: Levothyroxin

INTERVENTIONS:
Drug: Levothyroxin — Single-dose administration of 600 mcg of Levothyroxin for the assessment of bioequivalence
  Other Names: BC-T4CYS 150 µg tablet (Berlin-Chemie AG)
  Arms: BC-T4CYS 150 µg tablet (Berlin-Chemie AG)
Drug: Levothyroxin — Single-dose administration of 600 mcg of Levothyroxin for the assessment of bioequivalence
  Other Names: Letrox® 150 µg tablet (Berlin-Chemie AG),
  Arms: Letrox® 150 µg tablet (Berlin-Chemie AG),

SUMMARY:
Levothyroxine-sodium Bioequivalence Trial With Oral Single Dose Administration

DETAILED DESCRIPTION:
Single centre, open-label, randomised (order of treatments), balanced, 2-period, 2-sequence, single dose cross-over trial with administrations under fasting conditions separated by a washout period of at least 45 treatment-free days

ELIGIBILITY:
Inclusion Criteria:

1. ethnic origin: Caucasian
2. age: 18 years or older
3. body-mass index (BMI): 18.5 kg/m² and 30.0 kg/m²
4. good state of health
5. non-smoker or ex-smoker for at least 3 months
6. written informed consent, must be signed and dated before enrolment by the subject and the (sub-)investigator, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

Subjects cannot be included if they match any of the following exclusion criteria:

Safety concerns

1. existing cardiac, cardiovascular (e.g. angina pectoris, coronary heart disease) and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
2. existing hepatic and/or renal diseases and/or endocrine diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient
3. existing lipo-metabolic disorder or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient
4. existing gastrointestinal diseases or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
5. any disorder of thyroid glands reported in medical history resulting in an impairment of thyroid functions
6. existing diabetes mellitus
7. current treatment with anticoagulant drugs
8. history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
9. existing epilepsy or current treatment with antiepileptic drugs
10. subjects with pulmonary diseases (bronchial asthma, bronchitis, COPD) or known respiratory depression
11. known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations
12. history of significant drug allergy (especially hypersensitivity to levothyroxine-sodium)
13. subjects with severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
14. systolic blood pressure < 90 or > 139 mmHg
15. diastolic blood pressure < 60 or > 89 mmHg
16. heart rate < 50 bpm or > 90 bpm
17. QTc interval > 450 ms for men and > 470 ms for women
18. laboratory values out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator
19. ASAT > 20 % ULN, ALAT > 10 % ULN, bilirubin > 20 % ULN (except in case of existing Morbus Gilbert-Meulengracht deduced from anamnesis/medical history) and creatinine > 0.1 mg/dL ULN (limit of > 0.1 mg/dL correspondents to of > 9 µmol/l ULN).
20. positive anti-HIV-test (if positive to be verified by western blot), HBs-AG-test or anti-HCV-test
21. diagnosis of COVID-19 within the last 4 weeks and persisting disease symptoms (e.g. fever, cough) within 14 days prior to individual enrolment of the subject
22. direct contact with insufficient protection to persons in foreign risk regions for COVID-19 as defined by the Robert Koch Institute within the last 14 days prior to individual enrolment of the subject
23. known direct contact with insufficient protection to persons with diagnosis of COVID-19 within the last 14 days prior to individual enrolment upon reporting of the subject Lack of suitability for the clinical trial
24. acute or chronic diseases which may interfere with the pharmacokinetics of the IMP
25. history of or current drug or alcohol dependence
26. positive alcohol, cotinine or drug test at screening examination
27. regular intake of alcoholic food or beverages of ≥ 24 g pure ethanol for male or ≥ 12 g pure ethanol for female per day
28. subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
29. regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
30. blood donation or other blood loss of more than 400 ml within the last 2 months prior to individual screening of the subject
31. administration of any investigational medicinal product during the last 2 months prior to individual screening of the subject
32. regular treatment with any systemically available medication (except hormonal contraceptives or common replacement therapy with estrogens). In case of treatment with hormonal contraceptives or common replacement therapy with estrogens, the treatment should have started at least 3 months prior to the first IMP administration and be regularly continued during the clinical trial.
33. current treatment with medication for malaria prophylaxis
34. subjects, who report a frequent occurrence of migraine attacks
35. radiography with contrast medium within the last 6 weeks prior to the first administration

For female subjects with childbearing potential only:

36. positive pregnancy test at screening examination 37. pregnant or lactating women 38. female subjects who do not agree to apply highly effective contraceptive methods (highly effective contraceptive methods are defined in chapter 13.2.1) Administrative reasons 39. employee or family member of the Sponsor or the involved contract research organisation (CRO) 40. vulnerable subject defined as a soldier, a subject kept in detention, a protected adult under guardianship/trusteeship or committed to an institution by governmental or juridical order 41. subjects suspected or known not to follow instructions 42. subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial 43. no suitable candidate in the opinion of the investigator

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
AUC0-72 | 72 days
  AUC0-72 of levothyroxine (baseline corrected) after each treatment
Cmax | 72 days
  Cmax of levothyroxine (baseline corrected) after each treatment

SECONDARY OUTCOMES:
AUC0-tlast | 72 days
  AUC0-tlast of levothyroxine (baseline corrected) after each treatment
AUC0-∞ | 72 days
  AUC0-∞ of levothyroxine (baseline corrected) after each treatment
AUCexpol% | 72 days
  AUCexpol% of levothyroxine (baseline corrected) after each treatment
tmax | 72 days
  tmax of levothyroxine (baseline corrected) after each treatment
t1/2 | 72 days
  t1/2 of levothyroxine (baseline corrected) after each treatment
λz | 72 days
  λz of levothyroxine (baseline corrected) after each treatment
tlag | 72 days
  tlag of levothyroxine (baseline corrected) after each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Warnke André, Dr., Study Director — SocraTec R&D GmbH
Locations (1):
- Phase I Unit, Erfurt, Thuringia, Germany